CLINICAL TRIAL: NCT02203916
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-491 in Korean Subjects With Essential Hypertension
Brief Title: Azilsartan Medoxomil (TAK-491) Compared to Placebo in Korean Adults With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491_307; U1111-1130-9186 (Other: WHO)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: Drug therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 40 mg (Experimental): Azilsartan medoxomil 40 mg, tablets, orally, once daily for 6 weeks.
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan Medoxomil 80 mg (Experimental): Azilsartan medoxomil 80 mg, tablets, orally, once daily for 6 weeks.
  Interventions: Drug: Azilsartan medoxomil
- Placebo (Placebo Comparator): Azilsartan medoxomil placebo-matching tablets, orally, once daily for 6 weeks.
  Interventions: Drug: Azilsartan medoxomil placebo

INTERVENTIONS:
Drug: Azilsartan medoxomil — Azilsartan medoxomil tablets
  Other Names: TAK-491
  Arms: Azilsartan Medoxomil 40 mg; Azilsartan Medoxomil 80 mg
Drug: Azilsartan medoxomil placebo — Azilsartan medoxomil placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the antihypertensive effect of azilsartan medoxomil versus placebo in Korean adults with essential hypertension.

DETAILED DESCRIPTION:
The drug being tested in this study is called azilsartan medoxomil. Azilsartan medoxomil is being tested to treat Korean adults with hypertension. This study will look at changes in blood pressure in people who take azilsartan medoxomil.

The study will enroll approximately 325 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Azilsartan medoxomil 40 mg
* Azilsartan medoxomil 80 mg
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take two tablets at the same time each day throughout the study.

This multi-centre trial will be conducted in Korea. The overall time to participate in this study is 12 weeks. Participants will make 7 visits to the clinic, and will be contacted by telephone 7 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative, signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is treated with antihypertensive therapy and has a post-washout mean sitting clinic systolic blood pressure (SBP) ≥150 and ≤180 mm Hg on Day 1; or the patient has not received antihypertensive treatment within 28 days prior to Screening and has a mean sitting clinic SBP ≥150 and ≤180 mm Hg at the Screening Visit and on Day 1.
4. Is male or female aged ≥19 years.
5. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent through 30 days after last study drug dose.
6. Is willing to discontinue current antihypertensive medications on Day -21. If on amlodipine or chlorthalidone prior to Screening, the participant is willing to discontinue this medication on Day -28.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received TAK-491 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has sitting trough clinic diastolic blood pressure (DBP) greater than 114 mm Hg at Day 1 (after placebo run-in).
5. Has a history of hypersensitivity to TAK-491 (azilsartan medoxomil), any of its excipients, or other angiotensin-converting enzyme (ARBs).
6. Has a history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
7. Has clinically significant cardiac conduction defects (e.g., 3rd degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation, or flutter).
8. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease and hypertrophic obstructive cardiomyopathy (HOCM).
9. Has secondary hypertension of any etiology (e.g., renovascular disease, pheochromocytoma, Cushing syndrome).
10. Is noncompliant (less than 70% or greater than 130%) with study medication during placebo run-in period.
11. Has severe renal dysfunction or disease (confirmed by calculated creatinine clearance <30 mL/min/1.73m^2) at Screening.
12. Has known or suspected unilateral or bilateral renal artery stenosis.
13. Has a history of drug or alcohol abuse within the past 2 years.
14. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those patients with basal cell or stage I squamous cell carcinoma of the skin.)
15. Has type 1 or poorly controlled type 2 diabetes mellitus (hemoglobin A1c [HbA1c]>8.0%) at Screening.
16. Has an alanine aminotransferase (ALT) level greater than 2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
17. Has hyperkalemia (defined as serum potassium greater than the upper limit of normal per the central laboratory) at Screening.
18. Has any other serious disease or condition at screening or randomization that would compromise participant safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
19. Is required to take excluded medications.
20. If female, is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (15):
- South Korea (15):
  - Chuncheon, Gangwon-do
  - Wŏnju, Gangwon-do
  - Anyang-si, Gyeonggi-do
  - Goyang-si, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Daegu, Gyeongsangbuk-do
  - Yangsan, Gyeongsangnam-do
  - Jeonju, Jeollabuk-do
  - Gwangju, Jeollanam-do
  - Busan
  - Daegu
  - Daejeon
  - Incheon
  - Seoul

REFERENCES:
- [Derived] Juhasz A, Wu J, Hisada M, Tsukada T, Jeong MH. Efficacy and safety of azilsartan medoxomil, an angiotensin receptor blocker, in Korean patients with essential hypertension. Clin Hypertens. 2018 Feb 7;24:2. doi: 10.1186/s40885-018-0086-4. eCollection 2018. PMID 29445520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 29 investigative sites in Korea from 12 July 2014 to 03 February 2016.
Pre-assignment Details: Participants with a diagnosis of essential hypertension were randomized at a ratio of 2:2:1 into 1 of 3 treatment groups, once a day azilsartan medoxomil 40 mg, 80 mg or placebo. One participant in the 80 mg group was randomized twice, counted once in the randomized set, and is excluded from the Full Analysis Set and Safety Analysis Set.
Period: Overall Study
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg
Started | 65 | 132 | 131 (1 participant was randomized twice and counted only once.)
Full Analysis Set (FAS) | 65 | 132 | 130 (1 participant was randomized twice, counted once in randomized set, and excluded from the FAS.)
Safety Analysis Set (SAS) | 65 | 132 | 130 (1 participant was randomized twice, counted once in randomized set, and excluded from the SAS.)
Completed | 57 | 122 | 120
Not Completed | 8 | 10 | 11
Not completed — Pretreatment Event/Adverse Event | 1 | 3 | 2
Not completed — Major Protocol Deviation | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Voluntary Withdrawal | 3 | 3 | 8
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Reason Not Specified | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who received at least 1 dose of double-blind study drug and were randomized only once.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Total
Number analyzed (Participants) | 65 | 132 | 130 | 327
Age, Continuous [Mean (Standard Deviation); unit: years]
  Overall Study | 58.8 (10.21) | 59.8 (10.75) | 58.3 (11.57) | 59.0 (10.97)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 37 | 37 | 88
  Male | 51 | 95 | 93 | 239
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 65 | 132 | 130 | 327
Region of Enrollment [Number; unit: participants]
  Korea, Republic Of | 65 | 132 | 130 | 327
Height [Mean (Standard Deviation); unit: cm] | 166.1 (8.43) | 164.8 (9.09) | 165.6 (8.00) | 165.4 (8.53)
Weight [Mean (Standard Deviation); unit: kg] | 70.85 (9.892) | 70.97 (12.636) | 70.32 (13.070) | 70.69 (12.291)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.64 (2.653) | 26.02 (3.272) | 25.50 (3.460) | 25.74 (3.237)
Smoking Classification [Number; unit: participants]
  Never smoked | 29 | 71 | 65 | 165
  Current smoker | 12 | 22 | 26 | 60
  Ex-smoker | 24 | 39 | 39 | 102
Female Reproductive Status [Number; unit: participants] — Female participants only (n=14, 37, 37)
  participants
    Postmenopausal | 9 | 28 | 24 | 61
    Surgically Sterile | 2 | 4 | 3 | 9
    Of Childbearing Potential | 3 | 5 | 10 | 18
Estimated Glomerular Filtration Rate(eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 85.72 (14.798) | 87.44 (18.393) | 88.68 (18.443) | 87.59 (17.740)
Diabetes Status [Number; unit: participants]
  Yes | 4 | 21 | 13 | 38
  No | 61 | 111 | 117 | 289

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Trough Clinic Sitting Systolic Blood Pressure (SBP)
Description: The change in trough clinic sitting systolic blood pressure measured at week 6 relative to baseline. The trough is the average of the non-missing values of 3 serial trough sitting systolic blood pressure measurements. Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 6 blood pressure was measured approximately 24 hours after the previous day's dose. An analysis of covariance (ANCOVA) model, with treatment group as a fixed effect and Baseline sitting clinic systolic blood pressure as a covariate was used for analysis.
Time Frame: Baseline and Week 6
Population: Participants from the Full Analysis Set (FAS), including all randomized participants, who received at least 1 dose of double-blind study drug, with both a Baseline value and at least 1 post-baseline value, who were randomized only once. Missing values were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg
Number analyzed (Participants) | 63 | 127 | 129
mmHg | -8.776 (2.0039) | -22.093 (1.4117) | -23.731 (1.4017)
Statistical Analysis 1: Comparison: Placebo vs Azilsartan Medoxomil 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Overall type 1 error rate of 0.05 was controlled using principle of 'closed' testing: each pairwise comparison to placebo was conducted at 0.05 level with no p-value adjustment if hypothesis "all treatment groups equal" was first rejected at 0.05; Post-baseline p-values were from an ANCOVA model with treatment as a fixed factor and baseline values as a continuous covariate; LS Mean Difference = -13.317, 95% CI 2-sided [-18.138 to -8.497], Standard Error of Mean 2.4502
Statistical Analysis 2: Comparison: Placebo vs Azilsartan Medoxomil 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -14.955, 95% CI 2-sided [-19.770 to -10.141], Standard Error of Mean 2.4470

2. Secondary Outcome: Change From Baseline to Week 6 in Trough Clinic Sitting Diastolic Blood Pressure (DBP)
Description: The change in trough clinic sitting diastolic blood pressure measured at week 6 relative to baseline. The trough is the average of the non-missing values of 3 serial trough sitting diastolic blood pressure measurements. Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 6 blood pressure was measured approximately 24 hours after the previous day's dose. An analysis of covariance (ANCOVA) model, with treatment group as a fixed effect and Baseline sitting clinic diastolic blood pressure as a covariate was used for analysis.
Time Frame: Baseline and Week 6
Population: Participants from the FAS, including all randomized participants, who received at least 1 dose of double-blind study drug, with both a Baseline value and at least 1 post-baseline value, who were randomized only once. Missing values were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg
Number analyzed (Participants) | 63 | 127 | 129
mmHg | -2.6 (8.60) | -10.7 (10.12) | -11.6 (10.12)

3. Secondary Outcome: Percentage of Participants Who Achieved a Clinic DBP Response at Week 6
Description: Clinic DBP response is defined as clinic DBP <90 mmHg and/or reduction of ≥10 mmHg from Baseline. DBP is the arithmetic mean of 3 serial diastolic blood pressure measurements.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg
Number analyzed (Participants) | 63 | 127 | 129
percentage of participants | 42.9 | 83.5 | 85.3

4. Secondary Outcome: Percentage of Participants Who Achieved a Clinic SBP Response at Week 6
Description: SBP response is defined as clinic SBP <140 mmHg and/or reduction of ≥20 mmHg from Baseline. SBP is the arithmetic mean of 3 serial systolic blood pressure measurements.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg
Number analyzed (Participants) | 63 | 127 | 129
percentage of participants | 38.1 | 63.0 | 65.9

5. Secondary Outcome: Percentage of Participants Who Achieved Both a Clinic DBP and SBP Response at Week 6
Description: Percentage of participants who achieved both a clinic DBP and SBP response measured at week 6 defined as clinic DBP <90 mmHg and/or reduction of ≥10 mmHg from Baseline AND clinic SBP <140 mmHg and/or reduction of ≥20 mmHg from Baseline. DBP and SBP are based on the arithmetic mean of 3 serial blood pressure measurements.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg
Number analyzed (Participants) | 63 | 127 | 129
percentage of participants | 25.4 | 62.2 | 65.9

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events: from the first dose of double-blind study drug to 14 days after the last dose (up to 66 days). Serious adverse events: from the first dose of double blind study drug to 30 days after the last dose (up to 82 days).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Data is presented for the Safety Analysis Set.
Arm/Group | Placebo | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/132 | 2/130
Other Adverse Events (participants affected / at risk) | 7/65 | 8/132 | 14/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Azilsartan Medoxomil 40 mg (N=132) | Azilsartan Medoxomil 80 mg (N=130)
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Azilsartan Medoxomil 40 mg (N=132) | Azilsartan Medoxomil 80 mg (N=130)
Dizziness (Nervous system disorders) | 0 | 3 | 7
Nasopharyngitis (Infections and infestations) | 3 | 2 | 4
Headache (Nervous system disorders) | 2 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.